CLINICAL TRIAL: NCT05161013
Title: A Proof-of-Concept Study Evaluating LINFU™: A Noninvasive Method for Increasing Exfoliation of Pancreatic Ductal Cells Into the Pancreatic Fluid for the Early Detection of Pancreatic Ductal Adenocarcinoma (PDAC)
Brief Title: A Proof-of-Concept Study Evaluating LINFU™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adenocyte, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Adenocyte 111
Record Dates: First submitted 2021-11-21; First posted 2021-12-16 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-11

CONDITIONS: Pancreas Adenocarcinoma; Dysplasia
Keywords: Pancreatic Neoplasm; Pancreatic Cancer; Early detection
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients at high risk of developing pancreatic cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- The LINFU™ test (Experimental): LINFU™ to increase sensitivity of pancreatic juice cytology LINFU™ consists of analysis of pancreatic fluid collected with the help of low intensity non-focused ultrasound excitation of the pancreas. Lumason, will be used to create bubbles and possibly increase the number of pancreatic cell we collect for the study. Secretin is also used to increase the number of pancreatic cell excretion to maximize the number of cells collected.
  Interventions: Diagnostic Test: LINFU™

INTERVENTIONS:
Diagnostic Test: LINFU™ — A method to detect pancreatic cancer (ductal adenocarcinoma) using ultrasound technology in those who are at significantly increased risk for developing pancreatic cancer. LINFU™ involves analysis of pancreatic fluid collected.

SUMMARY:
The purpose of this research study is to study a method to detect pancreatic precancer and cancer (ductal adenocarcinoma) using ultrasound technology in those who are at significantly increased risk for developing pancreatic cancer. The LINFU™ Technique is done by analysis of pancreatic fluid collected with the help of ultrasound. This is an investigational way to detect pancreatic precancers and ductal adenocarcinoma.

DETAILED DESCRIPTION:
Patients will undergo collection of pancreatic fluid by the LINFU™ Technique as part of this study. This procedure takes about 30-45 minutes. The details for the procedure are listed below.

LINFU™ Technique

1. Once the participant is sedated or under anesthesia, low intensity non-focused ultrasound excitation of the pancreas will be implemented. This means the sound waves from the ultrasound on the top of the stomach will be used to stimulate the pancreas to release juice.
2. During the ultrasound, the Investigator will administer Lumason through a vein in the participant's arm (IV). Lumason is a contrast agent that was frequently used to create bubbles that allows a better visualization of images. In this study, Lumason will be used to create bubbles and possibly increase the number of pancreatic cells collected for the study.
3. After 25 minutes of ultrasound, the participant will receive an IV dose of secretin over 1 minute. Naturally, secretin is a hormone released into the bloodstream by a part of the small intestine, namely duodenum, (especially in response to acidity) to stimulate secretion by the liver and pancreas. In this study, Secretin is used to increase the number of pancreatic cell excretion to maximize the number of cells collected.
4. The participant will then undergo EGD (insertion of a tube down the throat and past the stomach). EGD stands for esophagogastroduodenoscopy. The Investigator who is doing EGD will discuss all risks and explain how the procedure will be done.
5. The pancreatic juice will be collected immediately. About 15 minutes after the EGD procedure has begun, a second dose of secretin will be administered.
6. The pancreatic juice will continue to be collected for a total of 30 minutes.

The results of the LINFU technique will be provided to the investigator to help guide medical care. This is an experimental technique so participants won't receive the results. Participants will undergo clinical diagnostic procedures including EUS (endoscopic ultrasound) and/or MRI as part of the standard medical care and evaluation for pancreatic cancer. These procedures are not part of the study and the Investigator has already determined that these tests are required.

Participants will be called 24 hours after the study procedure and 30 days after the procedure to see if any symptoms of pancreatitis (inflammation of the pancreas have developed). If so, participants will be asked to come back to the clinic for further evaluation as would be done as part of the standard medical care. In addition, participants will have blood tests before the LINFU procedure and this will be repeated 24hours after the procedure. The blood tests will measure lipase levels to make sure there was no injury to the pancreas.

Any identifiable private information or specimens collected and/or used for the purposes of this research will not be used or distributed for future research studies.

ELIGIBILITY:
Inclusion criteria

1. Both males and females will be enrolled and must be at least 18 years of age and under age of 90
2. Patients at high risk of developing a pancreatic malignancy.
3. Patients undergoing EUS or receiving an MRI scan as part of their screening.
4. Institutional Review Board (IRB)-approved consent must be signed by patients to participate in this study.

Exclusion criteria

1. Patient under the age of 18 and over the age 90
2. Patients undergoing FNA
3. Contraindications to EUS as determined by study investigators.

   1. Patient with uncorrectable coagulopathy
   2. Patient that cannot undergo anesthesia due to cardio- pulmonary contraindication as deemed by the anesthesiologist
4. Patients undergoing EUS or ERCP for a suspected bile duct cancer arising from the intrahepatic or extrahepatic biliary epithelium
5. Pregnant females will be excluded.
6. Patient that is unable to provide informed consent
7. Patient with known allergy to Lumason or Secretin
8. Patients with an elevated baseline lipase level

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Does LINFU™ yield an adequate number of cells that can be used to help diagnose pancreatic precancers and cancers? | 4 months
  The cells obtained from all 10 patients undergoing LINFU™ will be analyzed microscopically and counted by a pathologist for adequacy of pancreatic cellular yield. For a LINFU test to be considered adequate, 100 well-preserved ductal cells per patient must be counted under the microscope. Cellularity of >50 or <100 cells per patient would be interpreted as "limited but adequate" and cellularity <50 cells is unsatisfactory for adequacy.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Corbett, MD, FASGE, Principal Investigator — Suncoast Endoscopy of Sarasota (a division of Florida Digestive Health Specialists)
Locations (1):
- Gastroenterology Associates of Sarasota, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No